CLINICAL TRIAL: NCT00499616
Title: Response- and Biology-Based Therapy for Intermediate-Risk Neuroblastoma
Brief Title: Combination Chemotherapy and Surgery With or Without Isotretinoin in Treating Young Patients With Neuroblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANBL0531; COG-ANBL0531 (Other: Children's Oncology Group); NCI-2009-00400 (Other: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Neuroblastoma
Keywords: regional neuroblastoma; disseminated neuroblastoma; stage 4S neuroblastoma; localized unresectable neuroblastoma; localized resectable neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Carboplatin; Cyclophosphamide; Doxorubicin; Etoposide; Topotecan; Isotretinoin; Surgical Procedures, Operative; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 2 (chemotherapy, surgery) (Experimental): 2 courses of initial chemotherapy (6 wks) - carboplatin, cyclophosphamide, doxorubicin hydrochloride, etoposide, filgrastim. Partial response (PR) to chemo go to observation. No PR: 2-6 additional courses of chemo (beginning course 3 - cyclophosphamide, etoposide, filgrastim, carboplatin, doxorubicin hydrochloride). No PR after additional chemotherapy proceed to retrieval chemo: cyclophosphamide and topotecan hydrochloride on days 1-5. Treatment with retrieval chemotherapy repeats every 21 days for up to 6 courses. Some patients may also undergo surgery.
  Interventions: Drug: carboplatin; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: topotecan hydrochloride; Procedure: Surgery; Drug: Filgrastim
- Group 3 (chemotherapy, surgery) (Experimental): 4 courses of initial chemo - carboplatin, cyclophosphamide, doxorubicin hydrochloride, filgrastim. Patients with a PR after chemo proceed to observation. No PR receive 2-4 additional courses of chemotherapy (beginning with course 5) - carboplatin, cyclophosphamide, doxorubicin hydrochloride, etoposide, filgrastim. No PR after additional chemo proceed to retrieval chemo - cyclophosphamide and topotecan hydrochloride. Some patients may also undergo surgery.
  Interventions: Drug: carboplatin; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: topotecan hydrochloride; Procedure: Surgery; Drug: Filgrastim
- Group 4 (chemotherapy, surgery, antineoplastic therapy) (Experimental): 8 courses of initial chemo - carboplatin, cyclophosphamide, doxorubicin hydrochloride, etoposide, filgrastim. Patients < 12 months of age with stg 3, 4, or 4S (not including liver metastases) disease who achieve a very good PR (VGPR) to chemo proceed to observation. Patients 12-18 months of age with stg 3 or 4 who achieve VGPR proceed to isotretinoin therapy. No VGPR proceed to retrieval chemo - cyclophosphamide and topotecan hydrochloride. Some patients may also undergo surgery.
  Interventions: Drug: carboplatin; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: topotecan hydrochloride; Drug: Isotretinoin; Procedure: Surgery; Drug: Filgrastim
- Non-intermediate risk enrolled on intermediate risk trial (Experimental): The no treatment group assignment patients may have received some treatment on ANBL0531 but they were not evaluable on this study due to being non-intermediate risk and hence did not receive a treatment assignment on ANBL0531.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Drug: carboplatin — Given IV
  Other Names: Paraplatin; NSC #241240
  Arms: Group 2 (chemotherapy, surgery); Group 3 (chemotherapy, surgery); Group 4 (chemotherapy, surgery, antineoplastic therapy)
Drug: cyclophosphamide — Given IV
  Other Names: Cytoxan; NSC #26271
  Arms: Group 2 (chemotherapy, surgery); Group 3 (chemotherapy, surgery); Group 4 (chemotherapy, surgery, antineoplastic therapy)
Drug: doxorubicin hydrochloride — Given IV
  Other Names: Adriamycin; NSC #123127
  Arms: Group 2 (chemotherapy, surgery); Group 3 (chemotherapy, surgery); Group 4 (chemotherapy, surgery, antineoplastic therapy)
Drug: etoposide — Given orally
  Other Names: VePesid; VP-16; NSC #141540
  Arms: Group 2 (chemotherapy, surgery); Group 3 (chemotherapy, surgery); Group 4 (chemotherapy, surgery, antineoplastic therapy)
Drug: topotecan hydrochloride — Given IV
  Other Names: SKF-104864; Hycamtin; NSC #60969
  Arms: Group 2 (chemotherapy, surgery); Group 3 (chemotherapy, surgery); Group 4 (chemotherapy, surgery, antineoplastic therapy)
Drug: Isotretinoin — Given orally
  Other Names: 13-cis-retinoic acid; RO-43; 780; Accutane; Amnesteem; Claravis; Sotret; NSC#329481
  Arms: Group 4 (chemotherapy, surgery, antineoplastic therapy)
Procedure: Surgery — With the exception of patients with INSS 4S disease, patients undergo surgery to remove as much of the primary tumor and involved lymph nodes as can safely be accomplished.
Drug: Filgrastim — Administered subcutaneously or by IV beginning 24-48 hrs after the last dose of chemotherapy & continuing daily until the ANC is greater than or equal to 1500 following the myelosuppressive nadir . Supportive care given to stimulate neutrophil recovery following chemotherapy and to shorten the duration of chemotherapy-induced neutropenia. On ANBL0531 the use of filgrastim was required for patients less than 60 days of age and was optional for other patients.
  Other Names: Granulocyte Colony-Stimulating Factor, r-metHuG-CSF, G-CSF, Neupogen, NSC #614629
  Arms: Group 2 (chemotherapy, surgery); Group 3 (chemotherapy, surgery); Group 4 (chemotherapy, surgery, antineoplastic therapy)

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin, cyclophosphamide, etoposide, and doxorubicin hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Isotretinoin may help neuroblastoma cells become more like normal cells, and grow and spread more slowly. Giving combination chemotherapy before surgery may make the tumor smaller and make it more likely that the tumor can be surgically removed. It is not yet known what is the minimal amount of chemotherapy needed to achieve sufficient tumor shrinkage to control intermediate risk neuroblastoma and prevent tumor recurrence or metastases.

PURPOSE: This phase III trial is designed to reduce therapy for patients with favorable biology intermediate risk neuroblastoma by decreasing the number of chemotherapy cycles administered and by allowing for up to 50% residual tumor volume for patients with localized disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Reduce therapy for patients with intermediate-risk neuroblastoma while maintaining a 3-year overall survival (OS) rate of ≥ 95% by using a response-based duration of therapy algorithm.
* Maintain an overall 3-year OS rate of ≥ 90% for patients within each group.
* Utilize loss of heterozygosity, prospectively, at 1p36 and 11q23 to refine risk-stratification and treatment assignment, allowing patients whose tumors lack these chromosomal abnormalities to receive a reduction in therapy, and compare the outcome with patients treated on COG-A3961.
* Reduce intensity of therapy for patients 365 to < 547 days (12-18 months) of age with stage 4 neuroblastoma and favorable biological features and maintain a 3-year event-free survival (EFS) rate consistent with that for patients < 1 year of age with stage 4 neuroblastoma treated on COG-A3961.
* Reduce intensity of therapy for patients 365 to < 547 days (12-18 months) of age with stage 3 MYCN-nonamplified but unfavorable histology neuroblastoma and maintain a 3-year EFS rate consistent with that for patients < 1 year of age with stage 3, MYCN-nonamplified, unfavorable histology neuroblastoma treated on COG-A3961.
* Reduce surgical morbidity for patients with stage 4S neuroblastoma by allowing for biopsy only, rather than complete surgical resection, of the primary tumor.
* Systematically study the outcome of patients with stage 4S neuroblastoma who are unable to undergo biopsy for biology-based risk assignment.
* Determine if the extent of surgical resection correlates with the maintenance of local control, EFS and/or OS rates, and surgical complication rate.

Secondary

* Determine the results of a standard retrieval approach for patients with residual disease after 8 courses of initial therapy.
* Determine the results of a standard retrieval approach for patients with progressive, nonmetastatic disease.
* Identify additional biological surrogate markers for disease relapse and/or metastatic progression.
* Describe the neurologic outcome of patients with paraspinal neuroblastoma primary tumors.
* Correlate surgical biopsy technique with adequacy of tissue acquisition for biologic studies and with complications associated with the biopsy procedure.
* Prospectively validate the prognostic ability of the International Neuroblastoma Risk Group image-defined risk factor system, and compare the institutional assessment of image-defined risk factors with that of central review.

OUTLINE: This is a multicenter study. Patients are assigned to 1 of 3 treatment groups by risk-stratification based on age, stage (INSS stage 2, 3, 4, or 4S), MYCN status (amplified vs not amplified), histopathologic classification, tumor DNA index, and allelic status at chromosome bands 11q23 and 1p36.

* Initial chemotherapy: Courses of initial chemotherapy are administered every 21 days according to group assignment as outlined below:

  * Course 1: Patients receive carboplatin IV over 1 hour on day 1 and etoposide IV over 1 hour on days 1-3.
  * Course 2: Patients receive carboplatin IV over 1 hour, cyclophosphamide IV over 1 hour, and doxorubicin hydrochloride IV over 15 minutes on day 1.
  * Course 3: Patients receive cyclophosphamide IV over 1 hour on day 1 and etoposide IV over 1 hour on days 1-3.
  * Course 4: Patients receive carboplatin IV over 1 hour and doxorubicin hydrochloride IV over 15 minutes on day 1 and etoposide IV over 1 hour on days 1-3.
  * Course 5: Patients receive cyclophosphamide IV over 1 hour on day 1 and etoposide IV over 1 hour on days 1-3.
  * Course 6: Patients receive carboplatin IV over 1 hour, cyclophosphamide IV over 1 hour, and doxorubicin hydrochloride IV over 15 minutes on day 1.
  * Course 7: Patients receive carboplatin IV over 1 hour on day 1 and etoposide IV over 1 hour on days 1-3.
  * Course 8: Patients receive cyclophosphamide IV over 1 hour and doxorubicin hydrochloride IV over 15 minutes on day 1.

    * Group 2: Patients receive 2 courses of initial chemotherapy. Patients with a partial response (PR) (50-90% reduction in volume) to chemotherapy proceed to observation. Patients without a PR receive 2-6 additional courses of chemotherapy (beginning with course 3). Patients who do not achieve a PR after additional chemotherapy proceed to retrieval chemotherapy.
    * Group 3: Patients receive 4 courses of initial chemotherapy. Patients with a PR after chemotherapy proceed to observation. Patients without a PR receive 2-4 additional courses of chemotherapy (beginning with course 5). Patients who do not achieve a PR after additional chemotherapy proceed to retrieval chemotherapy.
    * Group 4: Patients receive 8 courses of initial chemotherapy. Patients under 12 months of age with stage 3, 4, or 4S disease who achieve a very good PR (VGPR) (> 90% reduction in the volume of the primary tumor and resolution of metastatic disease, with the exception of liver and skin metastases) to chemotherapy proceed to observation. Patients 12-18 months of age with stage 3 or 4 disease [age 365 to < 547 days at diagnosis, INSS stage 3, MYCN-NA, unfavorable histology, any ploidy and patients age 365 to < 547 days at diagnosis, INSS stage 4, MYCN-NA, favorable histology, DI > 1] who achieve a VGPR proceed to isotretinoin therapy. Patients who do not achieve a VGPR after 8 courses of initial chemotherapy +/- surgery will proceed to retrieval chemotherapy with cyclophosphamide/topotecan for 2-6 courses until a VGPR can be achieved with a combination of chemotherapy and surgery.
* Retrieval chemotherapy*: Patients receive cyclophosphamide IV over 30 minutes and topotecan IV over 30 minutes on days 1-5. Treatment repeats every 21 days for up to 6 courses.

  * Groups 2 and 3: Patients with a PR after 2-6 courses of retrieval chemotherapy proceed to observation. Patients without a PR after 2-6 courses of retrieval chemotherapy are removed from protocol therapy.
  * Group 4: Patients under 12 months of age with stage 4 disease with a VGPR after retrieval chemotherapy proceed to observation. Patients 12-18 months of age with stage 3 or 4 disease who achieve a VGPR after retrieval chemotherapy proceed to isotretinoin therapy. Patients who do not achieve a VGPR after retrieval chemotherapy are removed from protocol therapy.

Group 4 patients who develop progressive, non-metastatic disease within 3 years of study enrollment will also receive retrieval chemotherapy with cyclophosphamide and topotecan.

NOTE: *Patients who have previously received cyclophosphamide and topotecan to achieve first PR/VGPR are not eligible for this Retrieval Therapy.

* Surgery: With the exception of patients with INSS 4S disease, patients undergo surgery to remove as much of the primary tumor and involved lymph nodes as can safely be accomplished. Reassessment for definitive surgery (for patients who undergo biopsy only or partial resection at diagnosis) is made at the completion of scheduled chemotherapy (after course 2 for group 2, after course 4 for group 3, and after course 8 for group 4).
* Isotretinoin therapy: Beginning 3-4 weeks after completion of chemotherapy or 2 weeks post-operatively (for patients who undergo surgical resection), patients receive oral isotretinoin twice daily on days 1-14. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up periodically for up to 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed neuroblastoma, ganglioneuroblastoma, or ganglioneuroma/maturing subtype

  * Newly diagnosed disease
  * Intermediate-risk disease
  * Needle biopsies or involved bone marrow are not sufficient for INPC histologic classification
* Meets 1 of the following criteria:

  * Group 2

    * International Neuroblastoma Staging System (INSS) stage 2A/2B; < 50% resected or biopsy only; ≤ 12 years of age; MYCN-not amplified (NA); any histology and ploidy; normal 1p and 11q
    * INSS stage 3; age < 365 days; MYCN-NA; favorable histology (FH); hyperdiploid (DI) > 1; normal 1p and 11q
    * INSS stage 3; 365 days to 12 years of age; MYCN-NA; FH; normal 1p and 11q
    * INSS stage 4S; age < 365 days; MYCN-NA; FH; DI >1; normal 1p and 11q; clinically symptomatic
  * Group 3

    * INSS stage 2A/2B; < 50% resected or biopsy only; ≤ 12 years of age; MYCN-NA; any histology and ploidy; 1p loss of heterozygosity (LOH) and/or unb11q LOH (or data missing for either)
    * INSS stage 3; age < 365 days; MYCN-NA; FH; DI > 1; 1p LOH and/or unb11q LOH (or data missing for either)
    * INSS stage 3; age < 365 days; MYCN-NA; DI = 1 and/or unfavorable histology (UH); normal 1p and 11q
    * INSS stage 3; 365 days to 12 years of age; MYCN-NA; FH; 1p LOH and/or unb11q LOH (or data missing for either)
    * INSS stage 4; age < 365 days; MYCN-NA; FH; DI > 1; normal 1p and 11q
    * INSS stage 4S; age < 365 days; MYCN-NA; either UH and any ploidy or FH and DI = 1; normal 1p and 11q
    * INSS stage 4S; age < 365 days; MYCN-NA; FH; DI > 1; 1p LOH and/or unb11q LOH (or data missing for either); clinically symptomatic
  * Group 4

    * INSS stage 3; age < 365 days; MYCN-NA; DI = 1 and/or UH; 1p LOH and/or unb11q LOH (or data missing for either)
    * INSS stage 3; age 365 to < 547 days; MYCN-NA; UH; any ploidy; any 1p and 11q
    * INSS stage 4, age < 365 days; MYCN-NA; DI = 1 and/or UH; any 1p and 11q
    * INSS stage 4; age < 365 days; MYCN-NA; FH; DI > 1; 1p LOH and/or unb11q LOH (or data missing for either)
    * INSS stage 4; age 365 to < 547 days; MYCN-NA; FH; DI > 1; any 1p and 11q
    * INSS stage 4S; age < 365 days; MYCN-NA; UH and any ploidy or FH and DI = 1; 1p LOH and/or unb11q LOH (or data missing for either)
    * INSS stage 4S; age < 365 days; unknown or incomplete biologic features

      8 courses of initial chemo - carboplatin, cyclophosphamide, doxorubicin hydrochloride, etoposide, filgrastim.

Patients < 12 months of age with stg 3, 4, or 4S disease who achieve a very good PR (VGPR) to chemo (with the exception of resolution of skin or liver metastases in stage 4S patients) proceed to observation. Patients 12-18 months of age with stg 3 or 4 who achieve VGPR proceed to isotretinoin therapy. No VGPR proceed to retrieval chemo - cyclophosphamide and topotecan hydrochloride. Some patients may also undergo surgery.

* Must already be enrolled on protocol COG-ANBL00B1

  * Simultaneous enrollment on COG-ANBL00B1 and this study allowed for clinical situations in which emergent treatment may be indicated including, but not limited to, the following criteria:

    * Epidural or intraspinal tumors with existing or impending neurologic impairment
    * Periorbital or calvarial-based lesions with existing or impending cranial nerve impairment
    * Anatomic or mechanical compromise of critical organ function by tumor (e.g., abdominal compartment syndrome, urinary obstruction)
    * Asymptomatic but, in the opinion of the treating physician, it is in the patient's best interest to begin chemotherapy immediately due to impending risk of neurologic impairment or organ dysfunction
* If patient receives study chemotherapy prior to undergoing diagnostic biopsy, the biopsy must be performed within 96 hours of beginning study therapy

  * The only exception to this requirement is for patients with stage 4S disease who are considered too ill to undergo a diagnostic procedure will be waived the requirement for diagnostic tissue submission but will still need to be enrolled on COG-ANBL00B1

    * For patients with stage 4S disease who are very ill and in whom an open biopsy to obtain tissue for diagnosis and biologic studies is considered medically contraindicated, every effort should be made to obtain some tumor tissue by either fine-needle aspiration of a metastatic site of disease and/or sampling of involved bone marrow, so that this tumor sample can be submitted for MYCN determination
* Patients who require emergent therapy, either prior to the diagnostic biopsy or before biology features are available, can be enrolled simultaneously on COG-ANBL00B1 and COG-ANBL0531 to receive emergent protocol therapy

  * In emergent circumstances, COG-ANBL0531 protocol therapy may be initiated prior to enrollment on study as long as the patient has neuroblastoma by clinical diagnosis, all other COG-ANBL0531 eligibility criteria are met, and the COG-ANBL0531 Initial Therapy consent has been signed prior to starting protocol therapy; in this circumstance ANBL0531 enrollment must occur within 4 working days of starting protocol therapy
  * Clinical situations in which emergent enrollment and treatment may be indicated include, but are not limited to, the following circumstances:

    * Epidural or intraspinal tumors with existing or impending neurologic impairment
    * Periorbital or calvarial-based lesions with existing or impending cranial nerve impairment
    * Anatomic or mechanical compromise of critical organ function by tumor (e.g., abdominal compartment syndrome, urinary obstruction)
    * Evolving hepatomegaly in infants less than 2 months of age

PATIENT CHARACTERISTICS:

* See Disease Characteristics

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No other prior chemotherapy or radiotherapy with the exception of dexamethasone
* No participation in another COG study with tumor therapeutic intent

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 464 (Actual)
Dates: Start 2007-10-08 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clare Twist, MD, Study Chair — Lucile Packard Children's Hospital at Stanford University Medical Center; Mary Lou Schmidt, MD, Study Chair — University of Illinois at Chicago
Locations (189):
- United States (166):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children's Hospital Center for Cancer and Blood Disorders, Aurora, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Tripler AMC, Hawaii
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - University of Illinois Cancer Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Keyser Family Cancer Center at Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Simmons Cooper Cancer Institute, Springfield, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program at Barbara Bush Children's Hospital, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Floating Hospital for Children at Tufts - New England Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Children's Hospital, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Overlook Hospital, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center Hospital, Albany, New York
  - Maimonides Cancer Center at Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's - Dayton, Dayton, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - T.C. Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Carilion Medical Center for Children at Roanoke Community Hospital, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center - Tacoma, Tacoma, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center at Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (15):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Sainte Justine, Montreal, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen, Netherlands
- New Zealand (2):
  - Starship Children's Health, Auckland
  - Christchurch Hospital, Christchurch
- San Jorge Children's Hospital, Santurce, Puerto Rico

REFERENCES:
- [Derived] Twist CJ, Schmidt ML, Naranjo A, London WB, Tenney SC, Marachelian A, Shimada H, Collins MH, Esiashvili N, Adkins ES, Mattei P, Handler M, Katzenstein H, Attiyeh E, Hogarty MD, Gastier-Foster J, Wagner E, Matthay KK, Park JR, Maris JM, Cohn SL. Maintaining Outstanding Outcomes Using Response- and Biology-Based Therapy for Intermediate-Risk Neuroblastoma: A Report From the Children's Oncology Group Study ANBL0531. J Clin Oncol. 2019 Dec 1;37(34):3243-3255. doi: 10.1200/JCO.19.00919. Epub 2019 Aug 6. PMID 31386611
- [Derived] Twist CJ, Naranjo A, Schmidt ML, Tenney SC, Cohn SL, Meany HJ, Mattei P, Adkins ES, Shimada H, London WB, Park JR, Matthay KK, Maris JM. Defining Risk Factors for Chemotherapeutic Intervention in Infants With Stage 4S Neuroblastoma: A Report From Children's Oncology Group Study ANBL0531. J Clin Oncol. 2019 Jan 10;37(2):115-124. doi: 10.1200/JCO.18.00419. Epub 2018 Nov 16. PMID 30444686
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/
- See also: Maintaining Outstanding Outcomes Using Response- and Biology-Based Therapy for Intermediate-Risk Neuroblastoma: A Report From the Children's Oncology Group Study ANBL0531 — https://pubmed.ncbi.nlm.nih.gov/31386611/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 2 (Chemotherapy, Surgery) | Group 3 (Chemotherapy, Surgery) | Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy) | Non-intermediate Risk Enrolled on Intermediate Risk Trial
Started | 176 | 142 | 89 | 57
Completed | 161 | 114 | 53 | 0
Not Completed | 15 | 28 | 36 | 57
Not completed — Death | 1 | 5 | 3 | 1
Not completed — Lack of Efficacy | 5 | 0 | 19 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Physician Decision | 6 | 16 | 9 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Ineligible | 1 | 2 | 0 | 15
Not completed — Not evaluable | 0 | 0 | 0 | 41
Not completed — Patient/Parent Refusal | 1 | 5 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy): 8 courses of initial chemo - carboplatin, cyclophosphamide, doxorubicin hydrochloride, etoposide, filgrastim. Patients < 12 months of age with stg 3, 4, or 4S disease who achieve a very good PR (VGPR) to chemo (with the exception of resolution of skin or liver metastases in stage 4S patients) proceed to observation. Patients 12-18 months of age with stg 3 or 4 who achieve VGPR proceed to isotretinoin therapy. No VGPR proceed to retrieval chemo - cyclophosphamide and topotecan hydrochloride. Some patients may also undergo surgery.
- Total: Total of all reporting groups
Arm/Group | Group 2 (Chemotherapy, Surgery) | Group 3 (Chemotherapy, Surgery) | Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy) | Non-intermediate Risk Enrolled on Intermediate Risk Trial | Total
Number analyzed (Participants) | 176 | 142 | 89 | 57 | 464
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 176 | 142 | 89 | 57 | 464
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.23 (1.47) | .74 (.89) | .60 (.36) | 1.51 (1.83) | 0.99 (1.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 72 | 49 | 26 | 217
  Male | 106 | 70 | 40 | 31 | 247
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 26 | 7 | 6 | 57
  Not Hispanic or Latino | 150 | 109 | 74 | 49 | 382
  Unknown or Not Reported | 8 | 7 | 8 | 2 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 0 | 2
  Asian | 5 | 8 | 4 | 2 | 19
  Native Hawaiian or Other Pacific Islander | 3 | 4 | 0 | 1 | 8
  Black or African American | 23 | 12 | 8 | 9 | 52
  White | 133 | 92 | 59 | 40 | 324
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 12 | 26 | 16 | 5 | 59
Region of Enrollment [Number; unit: participants]
  New Zealand | 2 | 0 | 1 | 0 | 3
  Canada | 16 | 6 | 10 | 5 | 37
  United States | 153 | 131 | 78 | 50 | 412
  Australia | 5 | 5 | 0 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Rates
Description: OS time is calculated from date of enrollment until death, or until last contact if the patient is alive.
Time Frame: 3 years
Population: Eligible intermediate risk patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2 (Chemotherapy, Surgery) | Group 3 (Chemotherapy, Surgery) | Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy)
Number analyzed (Participants) | 175 | 140 | 89
percentage of participants | 99.4 [98.3 to 100.0] | 93.5 [89.4 to 97.7] | 88.4 [81.5 to 95.3]

2. Primary Outcome: Definitive Determination of the Prognostic Ability of 1p and 11q
Description: Addressed by a descriptive comparison of the EFS and OS rates for patients with 1p loss vs without 1p loss, and for those with unbalanced 11q vs normal 11q.
Time Frame: At baseline
Population: Eligible intermediate risk patients with 1p and 11q data.
Measure: Number (95% Confidence Interval); unit: percentage of 3 yr EFS/OS rate
Arm/Group | Group 2 (Chemotherapy, Surgery) | Group 3 (Chemotherapy, Surgery) | Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy)
Number analyzed (Participants) | 175 | 104 | 62
percentage of 3 yr EFS/OS rate
  EFS Eligible & evaluable patients without 1p loss: number analyzed (Participants) | 175 | 85 | 40
  EFS Eligible & evaluable patients without 1p loss | 87.2 [82.0 to 92.4] | 84.6 [76.8 to 92.5] | 65.4 [50.0 to 80.8]
  OS Eligible & evaluable patients without 1p loss: number analyzed (Participants) | 175 | 85 | 40
  OS Eligible & evaluable patients without 1p loss | 99.4 [98.3 to 100.0] | 92.8 [87.2 to 98.4] | 83.7 [71.6 to 95.8]
  EFS Eligible & evaluable patients with 1p loss: number analyzed (Participants) | 0 | 19 | 22
  EFS Eligible & evaluable patients with 1p loss |  | 94.7 [84.7 to 100.0] | 81.8 [65.2 to 98.4]
  OS Eligible & evaluable patients with 1p loss: number analyzed (Participants) | 0 | 19 | 22
  OS Eligible & evaluable patients with 1p loss |  | 94.7 [84.7 to 100.0] | 95.5 [86.5 to 100.0]
  EFS Eligible & evaluable patients with normal 11q: number analyzed (Participants) | 175 | 96 | 43
  EFS Eligible & evaluable patients with normal 11q | 87.2 [82.0 to 92.4] | 87.5 [80.7 to 94.2] | 73.3 [59.5 to 87.0]
  OS Eligible & evaluable patients with normal 11q: number analyzed (Participants) | 175 | 96 | 43
  OS Eligible & evaluable patients with normal 11q | 99.4 [98.3 to 100.0] | 93.7 [88.7 to 98.7] | 87.7 [77.4 to 98.1]
  EFS Eligible & evaluable patients w/unbalanced 11q: number analyzed (Participants) | 0 | 8 | 18
  EFS Eligible & evaluable patients w/unbalanced 11q |  | 75.0 [45.0 to 100.0] | 65.5 [42.7 to 88.2]
  OS Eligible & evaluable patients w/unbalanced 11q: number analyzed (Participants) | 0 | 8 | 18
  OS Eligible & evaluable patients w/unbalanced 11q |  | 87.5 [64.6 to 100.0] | 88.2 [72.9 to 100.0]

3. Primary Outcome: Comparison Between Reduce Intensity of Therapy for Patients With Stage 4 Neuroblastoma and Favorable Biological Features and Patients < 1 Year of Age With Stage 4 Neuroblastoma Treated on COG-A3961
Description: Addressed by the interim stopping rule and the comparison, by INSS stage, to the historical EFS rate of the analogous cohort of patients < 1 yrs of age.
Time Frame: Up to 3 years
Population: Eligible and evaluable patients with Stage 4 neuroblastoma, 12-18 months of age, and favorable biological features.
Measure: Number (95% Confidence Interval); unit: percentage of 3 yr EFS rate
Arm/Group | Group 3 (Chemotherapy, Surgery) | Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy)
Number analyzed (Participants) | 0 | 9
percentage of 3 yr EFS rate |  | 66.7 [35.9 to 97.5]
Statistical Analysis 1: Comparison: Group 3 (Chemotherapy, Surgery) vs Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy); The event-free survival distributions of patients between 12-18 months of age with Stage 4 neuroblastoma and favorable biological features on ANBL0531 and patients less than 12 months of age with Stage 4 neuroblastoma on A3961 were compared using the log-rank test; Test type: Other; p = .3212, Log Rank; Log Rank Test Statistic = .9841

4. Primary Outcome: Comparison Between Reduce Intensity of Therapy for Patients With Unfavorable Histology Neuroblastoma and Patients Unfavorable Histology Neuroblastoma Treated on COG-A3961
Description: as for outcome 3
Time Frame: Up to 3 years
Population: Eligible and evaluable patients with Stage 3 neuroblastoma, 12-18 months of age, MYCN non-amplified, and unfavorable histology.
Measure: Number; unit: percentage of 3 yr EFS rate
Arm/Group | Group 3 (Chemotherapy, Surgery) | Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy)
Number analyzed (Participants) | 0 | 2
percentage of 3 yr EFS rate |  | 100.0

5. Primary Outcome: Reduced Surgical Morbidity for Patients With Stage 4S Neuroblastoma
Description: Descriptive analyses of the proportion of stage 4S infants that experience a surgical or post-operative event.
Time Frame: Up to 3 years
Population: Eligible and evaluable patients with Stage 4S neuroblastoma that had a biopsy or resection.
Measure: Number (95% Confidence Interval); unit: Proportion
Arm/Group | Group 2 (Chemotherapy, Surgery) | Group 3 (Chemotherapy, Surgery) | Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy)
Number analyzed (Participants) | 17 | 19 | 7
Proportion | 0.18 [0.06 to 0.41] | 0.11 [0.03 to 0.31] | 0 [0 to 0]

6. Primary Outcome: Outcome of Patients With Stage 4S Neuroblastoma Who Are Unable to Undergo Biopsy for Biology-based Risk Assignment
Description: Kaplan-Meier curves and lifetables of Event Free Survival (EFS) and Overall Survival (OS) rates will be generated to describe the outcome of the stage 4S infants unable to undergo biopsy.
Time Frame: From baseline to up to 10 years
Population: Eligible and evaluable patients with Stage 4S neuroblastoma unable to undergo biopsy.
Measure: Number (95% Confidence Interval); unit: percentage survival
Arm/Group | Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy)
Number analyzed (Participants) | 4
percentage survival
  OS | 50.0 [1.0 to 99.0]
  EFS | 25.0 [0 to 67.4]

7. Primary Outcome: Correlation Between Extent of Surgical Resection With the Maintenance of Local Control, Event Free Survival (EFS)
Description: To test the predictive ability of the extent of surgical resection for EFS, log-rank tests will be performed comparing complete surgical resection vs. without complete surgical resection.
Time Frame: Up to 10 years
Population: Eligible and evaluable intermediate risk patients with reported surgery
Measure: Number (95% Confidence Interval); unit: percentage of 3 yr EFS survival
Arm/Group | Group 2 (Chemotherapy, Surgery) | Group 3 (Chemotherapy, Surgery) | Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy)
Number analyzed (Participants) | 174 | 137 | 81
percentage of 3 yr EFS survival
  EFS w/complete surgical resection: number analyzed (Participants) | 65 | 43 | 28
  EFS w/complete surgical resection | 95.4 [90.0 to 100.0] | 88.4 [78.7 to 98.1] | 78.6 [63.4 to 93.8]
  EFS w/o complete surgical resection: number analyzed (Participants) | 109 | 94 | 53
  EFS w/o complete surgical resection | 82.2 [74.6 to 89.8] | 85.1 [77.7 to 92.4] | 69.2 [56.3 to 82.1]
Statistical Analysis 1: Comparison: Group 2 (Chemotherapy, Surgery) vs Group 3 (Chemotherapy, Surgery) vs Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy); The event-free survival distributions of patients with complete surgical resection and patients without complete surgical resection were compared using the log-rank test; Test type: Other; p = .0253, Log Rank; Log-Rank Test Statistic = 5.0049

8. Primary Outcome: Correlation Between Extent of Surgical Resection With the Maintenance of Local Control, Overall Survival (OS) Rates
Description: To test the predictive ability of the extent of surgical resection for OS, log-rank tests will be performed comparing complete surgical resection vs. without complete surgical resection.
Time Frame: Up to 10 years
Population: Eligible and evaluable intermediate risk patients with reported surgery.
Measure: Number (95% Confidence Interval); unit: percentage of OS rate
Arm/Group | Group 2 (Chemotherapy, Surgery) | Group 3 (Chemotherapy, Surgery) | Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy)
Number analyzed (Participants) | 174 | 137 | 81
percentage of OS rate
  OS w/complete surgical resection: number analyzed (Participants) | 65 | 43 | 28
  OS w/complete surgical resection | 100.0 [100.0 to 100.0] | 95.4 [89.0 to 100.0] | 96.4 [89.4 to 100.0]
  OS w/o complete surgical resection: number analyzed (Participants) | 109 | 94 | 53
  OS w/o complete surgical resection | 99.1 [97.2 to 100.0] | 93.5 [88.4 to 98.6] | 86.5 [77.0 to 96.0]
Statistical Analysis 1: Comparison: Group 2 (Chemotherapy, Surgery) vs Group 3 (Chemotherapy, Surgery) vs Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy); Test type: Other — The overall survival distributions of patients with complete surgical resection and patients without complete surgical resection were compared using the log-rank test; p = .1022, Log Rank; Log Rank Test Statistic = 2.6709

9. Primary Outcome: Correlation Between Extent of Surgical Resection With the Maintenance of Local Control, Surgical Complication Rate
Description: To test for the association of the extent of surgical resection (CR vs <CR) with surgical complications rate (complications of any kind vs no complications at all), a chi-square test will be performed.
Time Frame: Up to 10 years
Population: Eligible and evaluable intermediate risk patients with reported surgery
Measure: Number (95% Confidence Interval); unit: Proportion with surgical complications
Arm/Group | Group 2 (Chemotherapy, Surgery) | Group 3 (Chemotherapy, Surgery) | Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy)
Number analyzed (Participants) | 174 | 137 | 81
Proportion with surgical complications
  CR with complications: number analyzed (Participants) | 65 | 43 | 28
  CR with complications | .32 [.22 to .44] | .19 [.10 to .33] | .18 [.08 to .36]
  CR with no complications: number analyzed (Participants) | 109 | 94 | 53
  CR with no complications | .14 [.09 to .21] | .13 [.07 to .21] | .09 [.04 to .20]
Statistical Analysis 1: Comparison: Group 2 (Chemotherapy, Surgery) vs Group 3 (Chemotherapy, Surgery) vs Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy); The association between extent of surgical resection with occurrence of complications was determined using the chi-square test; Test type: Other; p = .0016, Chi-squared; Chi-Square Test Statistic = 9.9111

10. Secondary Outcome: Second-event-free Survival (E2FS)
Description: E2FS (from time of first event) will be calculated to describe the outcome for patients who have a first progressive, non-metastatic event during Observation and then receive protocol retrieval therapy.
Time Frame: From the time of the first progressive, non-metastatic event until the subsequent occurrence of relapse, progressive disease, secondary malignancy, or death; up to 3 years
Population: Eligible patients who have a first progressive, non-metastatic event during Observation and then receive protocol retrieval therapy
Measure: Number (95% Confidence Interval); unit: Percentage
Groups:
- All Patients: All eligible patients who have a first progressive, non-metastatic event during Observation and then receive protocol retrieval therapy
Arm/Group | All Patients
Number analyzed (Participants) | 7
Percentage | 57.14 [20.49 to 93.79]

11. Secondary Outcome: Second-Overall Survival
Description: OS (from the time of first event) will be calculated to describe the outcome for patients who have a first progressive, non-metastatic event during Observation and then receive protocol retrieval therapy.
Time Frame: From the time of the first progressive, non-metastatic event; up to 3 years
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | All Patients
Number analyzed (Participants) | 7
Percentage | 85.71 [59.78 to 100]

12. Secondary Outcome: Biological Surrogate Markers
Description: Multivariable analyses will be performed to identify variables of prognostic interest.
Time Frame: At baseline and surgery
Population: The data was not collected to assess this study aim.
Arm/Group | Group 2 (Chemotherapy, Surgery) | Group 3 (Chemotherapy, Surgery) | Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy)
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Neurologic Symptoms
Description: Percentage of patients with neurologic symptoms will be calculated. Includes patients with paraspinal or intraspinal tumors, including epidural tumors with or without spinal cord compression. Neurologic symptoms include back or extremities neurologic symptoms, motor deficit, abnormal sensation, abnormal bladder/bowel sphincteric function, chronic pain in back or extremities, scoliosis, kyphosis, or clinically relevant/functional abnormality in size or contour of leg or foot.
Time Frame: At baseline
Population: All eligible and evaluable patients enrolled on ANBL0531
Measure: Number; unit: percentage of patients
Arm/Group | Group 2 (Chemotherapy, Surgery) | Group 3 (Chemotherapy, Surgery) | Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy)
Number analyzed (Participants) | 175 | 141 | 88
percentage of patients | 36.57 | 35.46 | 27.27

14. Secondary Outcome: Association Between Surgical Biopsy Technique With Adequacy of Tissue Acquisition for Biologic Studies, and With Complications Associated With the Biopsy Procedure
Description: A chi-square test will be performed.
Time Frame: During and after surgery
Population: The data was not collected to assess this study aim.
Arm/Group | Group 2 (Chemotherapy, Surgery) | Group 3 (Chemotherapy, Surgery) | Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy)
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Image Defined Risk Factor (IDRF)
Description: Percentage of patients with presence of one or more IDRFs will be calculated. IDRFs describe anatomic features which may make surgical resection more difficult.
Time Frame: At baseline
Population: All eligible and evaluable patients enrolled on ANBL0531
Measure: Number; unit: percentage of patients
Arm/Group | Group 2 (Chemotherapy, Surgery) | Group 3 (Chemotherapy, Surgery) | Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy)
Number analyzed (Participants) | 175 | 141 | 88
percentage of patients | 54.86 | 60.28 | 56.82

ADVERSE EVENTS:
Description: SAE field contains NCI CTCAEs submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs.
Arm/Group | Group 2 (Chemotherapy, Surgery) | Group 3 (Chemotherapy, Surgery) | Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy) | Non-intermediate Risk Enrolled on Intermediate Risk Trial
Serious Adverse Events (participants affected / at risk) | 2/175 | 5/140 | 8/89 | 1/42
Other Adverse Events (participants affected / at risk) | 135/175 | 114/140 | 76/89 | 23/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 2 (Chemotherapy, Surgery) (N=175) | Group 3 (Chemotherapy, Surgery) (N=140) | Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy) (N=89) | Non-intermediate Risk Enrolled on Intermediate Risk Trial (N=42)
13200-Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
46300-Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
24600-Death NOS (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
55700-Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
40600-Hepatobiliary disorders - Other specify (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
44800-Infections and infestations - Other specify (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
73700-Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
80700-Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
17400-Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
58300-Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
65800-Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
10700-Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
11100-Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
71000-Renal and urinary disorders - Other specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
19200-Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
43900-Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
71500-Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
71600-Respiratory thoracic and mediastinal disorders - Other specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
43600-Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 2 (Chemotherapy, Surgery) (N=175) | Group 3 (Chemotherapy, Surgery) (N=140) | Group 4 (Chemotherapy, Surgery, Antineoplastic Therapy) (N=89) | Non-intermediate Risk Enrolled on Intermediate Risk Trial (N=42)
13200-Anemia (Blood and lymphatic system disorders) | 60 (94) | 64 (102) | 45 (105) | 14 (14)
17200-Blood and lymphatic system disorders - Other specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
25800-Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
33300-Febrile neutropenia (Blood and lymphatic system disorders) | 24 (28) | 22 (27) | 17 (20) | 1 (1)
20000-Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
51700-Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
87100-Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
55000-Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
29200-Endocrine disorders - Other specify (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
31900-Eye disorders - Other specify (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
10100-Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
10300-Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
14900-Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
25700-Diarrhea (Gastrointestinal disorders) | 6 (6) | 4 (4) | 5 (10) | 2 (2)
27600-Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
36700-Gastrointestinal disorders - Other specify (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (5) | 0 (0)
37600-Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
44600-Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
46300-Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
49400-Jejunal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
53900-Malabsorption (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
55600-Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
57600-Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
75700-Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
75900-Small intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
81900-Typhlitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
87900-Vomiting (Gastrointestinal disorders) | 5 (5) | 3 (3) | 4 (4) | 1 (1)
28200-Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
28300-Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
28400-Edema trunk (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
33900-Fever (General disorders) | 2 (2) | 1 (1) | 4 (4) | 0 (0)
34600-Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
35000-Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
37200-General disorders and administration site conditions - Other specify (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
43700-Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
48700-Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
58600-Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
60600-Pain (General disorders) | 2 (2) | 3 (4) | 1 (1) | 1 (1)
35400-Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
40000-Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
66600-Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
13100-Anaphylaxis (Immune system disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
10200-Abdominal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
16600-Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
16800-Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
18800-Bronchial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
20500-Catheter related infection (Infections and infestations) | 3 (4) | 7 (7) | 6 (6) | 0 (0)
29500-Enterocolitis infectious (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
32000-Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
38300-Gum infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
44800-Infections and infestations - Other specify (Infections and infestations) | 32 (50) | 19 (26) | 34 (60) | 6 (9)
50300-Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
53100-Lung infection (Infections and infestations) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
60100-Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
69800-Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
72600-Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
75200-Skin infection (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
80900-Tracheitis (Infections and infestations) | 0 (0) | 3 (5) | 0 (0) | 1 (1)
82300-Upper respiratory infection (Infections and infestations) | 1 (1) | 2 (4) | 3 (3) | 0 (0)
83100-Urinary tract infection (Infections and infestations) | 5 (5) | 1 (1) | 4 (5) | 0 (0)
88900-Wound infection (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
14500-Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
86400-Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
10900-Activated partial thromboplastin time prolonged (Investigations) | 3 (3) | 4 (5) | 3 (3) | 1 (1)
11600-Alanine aminotransferase increased (Investigations) | 4 (4) | 7 (9) | 8 (11) | 1 (1)
11800-Alkaline phosphatase increased (Investigations) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
15000-Aspartate aminotransferase increased (Investigations) | 2 (2) | 8 (9) | 11 (14) | 4 (4)
17400-Blood bilirubin increased (Investigations) | 2 (2) | 10 (11) | 6 (7) | 2 (2)
34000-Fibrinogen decreased (Investigations) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
37500-GGT increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
45800-INR increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
52600-Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
53700-Lymphocyte count decreased (Investigations) | 11 (14) | 11 (11) | 14 (28) | 1 (1)
58300-Neutrophil count decreased (Investigations) | 99 (173) | 86 (178) | 55 (156) | 13 (13)
65800-Platelet count decreased (Investigations) | 57 (79) | 56 (85) | 40 (75) | 9 (9)
88300-Weight loss (Investigations) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
88500-White blood cell decreased (Investigations) | 47 (72) | 60 (89) | 36 (72) | 8 (8)
10700-Acidosis (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 0 (0) | 3 (3)
11900-Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
13500-Anorexia (Metabolism and nutrition disorders) | 8 (8) | 9 (16) | 4 (9) | 2 (2)
24700-Dehydration (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 5 (5) | 0 (0)
41300-Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 1 (1) | 3 (3)
41400-Hyperglycemia (Metabolism and nutrition disorders) | 6 (7) | 7 (7) | 3 (5) | 2 (2)
41600-Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5) | 1 (1) | 1 (1)
41700-Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
41800-Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
42500-Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
42600-Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (5) | 6 (7) | 6 (7) | 1 (1)
42700-Hypocalcemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 4 (4) | 2 (2)
42900-Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 3 (4) | 2 (2)
43100-Hypokalemia (Metabolism and nutrition disorders) | 8 (10) | 13 (15) | 15 (18) | 2 (2)
43300-Hyponatremia (Metabolism and nutrition disorders) | 6 (6) | 5 (5) | 6 (6) | 1 (1)
43500-Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
81700-Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
16200-Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
38700-Head soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
55900-Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
58000-Neoplasms benign malignant and unspecified (incl cysts and polyps) - Other specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
81800-Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
22000-Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
25300-Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
27700-Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
29000-Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
58100-Nervous system disorders - Other specify (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
63900-Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
64100-Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
70900-Recurrent laryngeal nerve palsy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
73600-Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
11100-Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
68300-Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
83000-Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
11300-Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
14100-Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
15100-Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
15400-Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
19200-Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
19300-Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
21900-Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
27800-Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
43900-Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5) | 2 (3) | 1 (1)
65900-Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
66300-Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
66400-Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
71600-Respiratory thoracic and mediastinal disorders - Other specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 2 (2) | 1 (1)
60800-Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
74700-Skin and subcutaneous tissue disorders - Other specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
84100-Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
19800-Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
39100-Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
42100-Hypertension (Vascular disorders) | 5 (6) | 2 (3) | 6 (15) | 1 (1)
43600-Hypotension (Vascular disorders) | 1 (2) | 3 (3) | 0 (0) | 3 (3)
53300-Lymph leakage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
79600-Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.